CLINICAL TRIAL: NCT05326854
Title: EVALUATION OF THE EFFECTIVENESS OF THE NAVIGATION ASSISTED CARE PROGRAM FOR WOMEN WITH MEDICAL TERMINATION
Brief Title: NAVIGATION ASSISTED CARE PROGRAM AND TERMINATION OF PREGNANCY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, havva yeşildere sağlam, Sub-Investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ESKISEHIROU1
Record Dates: First submitted 2022-03-18; First posted 2022-04-14 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Termination of Pregnancy; Supportive Care; Nursing Caries
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): 1., 2., 3. İnterview (in hospital) The patient will be educated. Measuring tools will be applied. (Personal Information Form- Coping and Adaptation Process Scale)( discharge: Perinatal Grief Scale, Depression Anxiety Stress Scale) The mobile application developed within the scope of post-termination support will be downloaded to the patient's phone. Informed consent form will be signed by the patient.
  Sharing problems, presenting solutions. Follow-up of the patient and strengthening and supporting in this process.
  4., 5., 6. Interview at home (following the patient with mobile application and phone calls)
  7. and 8., Interview at home (following the patient with mobile application and phone calls) Measuring tools will be appliedPerinatal Grief Scale, Depression, Anxiety and Stress Scale, Coping and Adaptation Process Scale
  Interventions: Other: supportive care
- Control Group (No Intervention): In the control group, data collection forms will be applied at admission and discharge to the service. There will be no application other than the routine care of the hospital. The routine care of the hospital applied to the control group within the scope of the research includes the information that should be given before, during and after the procedure that should be done depending on the medical intervention. In addition, there is no support program planned in the hospital and at discharge, and there is no follow-up after discharge.
  1. Interview at hospital Measuring tools will be applied Perinatal Grief Scale, Depression, Anxiety and Stress Scale, Coping and Adaptation Process Scale, Discharge time, labor pain.
  2. and 3. Interview at home Measuring tools will be applied Perinatal Grief Scale, Depression, Anxiety and Stress Scale, Coping and Adaptation Process Scale

INTERVENTIONS:
Other: supportive care — After Medical Termination Navigation Assisted Care Program admission to the service will be held in the form of three interviews in the clinic before and after termination. The planned training will be given in three sessions and a different training module will be applied in each meeting. After the patient is discharged, three sessions will be held remotely via telephone.
  Arms: intervention group

SUMMARY:
This study was planned to evaluate the effectiveness of the navigation-assisted care program based on the Swanson Theory of Care, which was developed for women who underwent medical termination as a result of a complication caused by maternal or fetal reasons.

DETAILED DESCRIPTION:
H1: Navigation-assisted care program based on Swanson care theory reduces perinatal grief levels of women.

H2: Navigation-assisted care program based on Swanson care theory reduces depression-anxiety-stress levels of women

H3: Navigation-assisted care program based on Swanson care theory positively affects women's coping and adjustment levels.

Independent variables: Sociodemographic characteristics such as age, marital status, educational status and the Navigation Assisted Care Program Based on Swanson Care Theory constitute the independent variables.

Dependent variables: Scores from Perinatal Grief Scale, Depression, Anxiety and Stress Scale, Coping and Adaptation Process Scale, discharge time, labor pain constitute the dependent variables.

Preparation of mobile application:

After the formation of the training content, expert opinions and the completion of the ethics committee process, the construction phase of the mobile application started. The mobile application was named "Pregnancy Loss Support Program". In order for the patients in the intervention group to log in to the mobile application, a user name and password were defined, and the user names and passwords defined during the installation of the mobile application were reported to them by the researcher. Before starting the patient interviews with the mobile application, trials were made and updates were made regarding the deficiencies. Continuous support was provided to people through the Messaging section, which offers instant messaging so that participants' questions can be answered. The questionnaires applied during the study were made available to the participants in the Survey section. In the video section, videos that will provide technical support for mobile application installation and use have been added. A symptom diary section was created in order for the participants to indicate the changes that occurred in them, and the participants were provided to report their symptoms from this section.

* After the patient is admitted to the service at the first interview, data collection forms will be applied to the women. Afterwards, information will be given about the mobile application and its use, and the mobile application will be downloaded to the women's phones. The mobile application will be activated after the discharge of the patient, and the woman will be able to access the mobile application at discharge. The mobile application will be installed on the patient's phone at the first meeting in the hospital, and the patient will be informed about its use.
* In the second meeting, before the termination, the Medical Post-Termination Training and Supportive Care Program will continue.
* After the termination at the third meeting, the Medical Post-Termination Training and Supportive Care Program will continue. Telephone interviews and follow-up plans will be made with the patient after discharge. After the medical termination decision is taken, it is thought that there may be deficiencies during the training due to the high anxiety and stress levels of women, and the training program will be integrated into the mobile application so that women can access it at any time. In case of a problem with the use of the mobile application, women will be able to reach the researcher by phone during working hours and support will be provided by the researcher. In the study, it was planned to make home visits, but the follow-ups arising from the Coronavirus Pandemic process will be made in the form of telephone follow-up and follow-up. Survey and measurement tools will be applied.(Perinatal Grief Scale, Depression, Anxiety and Stress Scale, Coping and Adaptation Process Scale)
* After the discharge, the fourth interview will take place in the first week, the problems experienced by the patient will be discussed and his questions will be answered. Post-Medical Termination Education and Supportive Care Program will continue.
* After discharge, the fifth interview will be held in the second week and the problems experienced by the patient will be discussed.
* After discharge, the sixth interview will be held in the fourth week and the problems experienced by the patient will be discussed.
* The seventh interview will be held in the sixth week after discharge, during which the problems experienced by the patient will be discussed, data collection forms and measurement tools will be applied. (Perinatal Grief Scale, Depression, Anxiety and Stress Scale, Coping and Adaptation Process Scale)
* The eighth interview will be held in the tenth week, during which the problems experienced by the patient will be discussed, data collection forms and measurement tools will be applied. (Perinatal Grief Scale, Depression, Anxiety and Stress Scale, Coping and Adaptation Process Scale)

Applications to the control group In the control group, data collection forms and measurement tools will be applied after admission to the service. No application will be made other than the routine maintenance of the hospital. The routine care of the hospital applied to the control group within the scope of the research includes the information that should be given before, during and after the procedure that should be done depending on the medical intervention. In addition, there is no support program planned in the hospital and at discharge, and there is no follow-up after discharge. In studies evaluating the effectiveness of education in the literature, 6-8 weeks are considered appropriate for evaluation. For this reason, the first measurement will be made in the 6th week of the study. In addition, in terms of evaluating the effects of medical termination on the woman in the long term, a post-test will be applied at the 10th week.

• After the completion of the training and evaluation in terms of ethical compliance, the support program training content and mobile application usage will be opened to the control group. Women in the control group will have access to the application after study protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Able to read and write,
* Agreeing to participate in the study,
* Accepting the decision of medical termination of pregnancy,
* Does not have a diagnosed psychiatric disease,
* Medical termination decision is taken in the first and second trimesters,
* Women who have a phone that can use the mobile application program will be included in the study.

Exclusion Criteria:

* Being under the age of 18,
* Those who do not agree to participate in the study,
* Women who do not have a phone that can use the mobile application program will not be included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
perinatal grief-1 | 2nd or 3rd days
  Evaluation will be made using the scale. Change will be evaluated at the after termination(birth) using the Perinatal grief scale
  Changes in the age of the patients over time will be evaluated. It will increase-decrease over time. The scale does not have any cutoff points. As the scale score increases, the level of grief increases
  The termination process of the patients may vary. The perinatal grief scale is first administered in the hospital after termination.
perinatal grief-2 | 8th weeks
  Evaluation will be made using the scale. Change will be evaluated at the 7th interview (at 6-8weeks) using the Perinatal grief scale
  Changes in the age of the patients over time will be evaluated. It will increase-decrease over time. The scale does not have any cutoff points. As the scale score increases, the level of grief increases
perinatal grief-3 | 12th weeks
  Evaluation will be made using the scale. Change will be evaluated at the 8th interview (at 10-12weeks) using the Perinatal grief scale
  Changes in the age of the patients over time will be evaluated. It will increase-decrease over time. The scale does not have any cutoff points. As the scale score increases, the level of grief increases
depression-anxiety-stress-1 | 2nd or 3rd days
  Change will be evaluated at the after termination(birth) using the Depression Anxiety Stress Scale-21.
  The depression anxiety stress scale is first interwiev in the hospital after termination. The patient is followed as long as he stays in the hospital.(avarage3-4 days) Depression anxiety stress level of the patients will be evaluated. Scale has certain cutoff points. Women's depression, anxiety and stress will be examined. Changes will be observed over time. Follow-up covers a period of 10-12 weeks. In this process, both follow-up and supportive care continue.
  Depression Anxiety Stress (Respectively) NORMAL 0-4 0-3 0-7 MILD 5-6 4-5 8-9 MEDİUM LEVEL 7-10 6-7 10-12 HIGH LEVEL 11-13 8-9 13-16 VERY HIGH 4+ 10+ 17+
depression-anxiety-stress-2 | 8th weeks
  Change will be evaluated at the 7th interview (at 6-8weeks using the Depression Anxiety Stress Scale-21.
  The depression anxiety stress scale is first interwiev in the hospital after termination. The patient is followed as long as he stays in the hospital.(avarage3-4 days) Depression anxiety stress level of the patients will be evaluated. Scale has certain cutoff points. Women's depression, anxiety and stress will be examined. Changes will be observed over time. Follow-up covers a period of 10-12 weeks. In this process, both follow-up and supportive care continue.
  Depression Anxiety Stress (Respectively) NORMAL 0-4 0-3 0-7 MILD 5-6 4-5 8-9 MEDİUM LEVEL 7-10 6-7 10-12 HIGH LEVEL 11-13 8-9 13-16 VERY HIGH 4+ 10+ 17+
depression-anxiety-stress-3 | 12th weeks
  Change will be evaluated at the 8th interview (at 10.-12weeks) using the Depression Anxiety Stress Scale-21.
  The depression anxiety stress scale is first interwiev in the hospital after termination. The patient is followed as long as she stays in the hospital.(avarage3-4 days) Depression anxiety stress level of the patients will be evaluated. Scale has certain cutoff points. Women's depression, anxiety and stress will be examined. Changes will be observed over time. Follow-up covers a period of 10-12 weeks. In this process, both follow-up and supportive care continue.
  Depression Anxiety Stress (Respectively) NORMAL 0-4 0-3 0-7 MILD 5-6 4-5 8-9 MEDİUM LEVEL 7-10 6-7 10-12 HIGH LEVEL 11-13 8-9 13-16 VERY HIGH 4+ 10+ 17+
coping and adaptation-1 | first day
  Evaluation will be made using the Coping and adaptation scale.
  Change will be evaluated in the hospital before termination(birth), using the Coping and Adaptation Process Scale
  The increase in the coping and adjustment levels of the patients will be evaluated.
  Follow-up covers a period of 10-12 weeks. In this process, both follow-up and supportive care continue.
  The Coping and Adaptation process scale, on the other hand, is first applied in the hospital after the hospitalization of the patients.
coping and adaptation-2 | 8th weeks
  Evaluation will be made using the scale. Coping and adaptation scale Change will be evaluated at the 7th interview (at 6-8weeks) using the Coping and Adaptation Process Scale
  The increase in the coping and adjustment levels of the patients will be evaluated.
  Follow-up covers a period of 10-12 weeks. In this process, both follow-up and supportive care continue.
coping and adaptation-3 | 12th weeks
  Evaluation will be made using the scale. Coping and adaptation scale Change will be evaluated at the 8th interview (at 10.-12weeks) using the Coping and Adaptation Process Scale
  The increase in the coping and adjustment levels of the patients will be evaluated.
  Follow-up covers a period of 10-12 weeks. In this process, both follow-up and supportive care continue.
Labor Pain-1 | first day
  Evaluation will be made using the VAS scale in hospital. The change in pain scores of the experimental group and the control group will be compared.
  1-The latent phase covers the period until the 3-4 cm gap in labor occurs. The pain he feels during this time will be measured with a visual analog scale.
  This process can take up to 1 day on average.
Labor Pain-2 | first day
  Evaluation will be made using the VAS scale in hospital. The change in pain scores of the experimental group and the control group will be compared.
  2-Pain during the act (baby's exit) will be measured with the visual analog scale.
  This process can take up to 1 day on average.
Labor Pain-3 | first day
  Evaluation will be made using the VAS scale in hospital. The change in pain scores of the experimental group and the control group will be compared.
  3-The pain felt by the baby for the first two hours after the action occurs will be measured with the visual analog scale.
  This process can take up to 1 day on average.

SECONDARY OUTCOMES:
discharge time | Avarage 3-4 days
  The length of stay in the hospital will be calculated. Time between hospitalization and discharge. (avarage3-4 days) The time spent in the hospital can last for 3-4 days on average.
quality of sleeping | 12th weeks
  Change will be evaluated at the 8th interview (at 10.-12weeks) using the VAS Scale.
  A high score from the scale indicates good sleep quality. There are no cutoff piont on the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Osmangazi Üniversitesi, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yesildere Saglam H, Gursoy E, Kartal Y. The effect of nursing care during pregnancy termination on women's prenatal grief, depression, anxiety, stress and coping levels: A randomized controlled study. Women Health. 2025 Jan;65(1):92-106. doi: 10.1080/03630242.2024.2441377. Epub 2024 Dec 18. PMID 39696803